CLINICAL TRIAL: NCT03823560
Title: Evaluation of Performance and Safety of the CE Marked Medical Device Class IIb Celegyn® in Vulvovaginal Atrophy (VVA): a Randomised, Double-blind, Parallel Groups, Multicentric, Placebo-Controlled, Prospective Clinical Study
Brief Title: Performance and Safety of Class IIb MD Celegyn® in VVA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nathura S.p.A (Industry)
Collaborators: Evidilya S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CeleMD01
Record Dates: First submitted 2019-01-23; First posted 2019-01-30 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Vulvovaginal Atrophy

STUDY DESIGN:
Intervention Model Description: randomised, double-blind, parallel groups, multicentric, placebo-controlled, prospective clinical study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP A: medical device Celegyn® (Experimental): Medical device Celegyn® presents itself as a white ivory cream (cream-like oil-in-water topical emulsion) with a typical smell; it is intended for topical use.
  Posology: It is to be applied preferably in the evening, once a day, for the first seven days, and every other day until the end of the study (i.e. during the second and third week) according to the following:
  * for external (vulvar) use: it should be applied as needed directly to the affected area with a gentle massage;
  * for internal (vaginal) use: use the vaginal applicators provided and follow the directions of use, according to package insert
  Interventions: Device: Celegyn®
- GROUP B: matching placebo (Placebo Comparator): Investigational Product (IP) placebo presents itself as a white ivory cream (cream-like oil-in-water topical emulsion) with a typical smell; it is intended for topical use.
  Posology: It is to be applied preferably in the evening, once a day, for the first seven days, and every other day until the end of the study (i.e. during the second and third week) according to the following:
  * for external (vulvar) use: it should be applied as needed directly to the affected area with a gentle massage;
  * for internal (vaginal) use: use the vaginal applicators provided and follow the directions of use, according to package insert
  Interventions: Device: Matching placebo

INTERVENTIONS:
Device: Celegyn® — Medical device Celegyn® presents itself as a cream.
  Arms: GROUP A: medical device Celegyn®
Device: Matching placebo — IP placebo presents itself as a cream.
  Arms: GROUP B: matching placebo

SUMMARY:
The aim of this study is primarily to investigate the performance of Celegyn®, a hyaluronic acid-based vaginal cream (CE marked 0546 medical device), enriched with plant-based ingredients, in comparison with placebo, in promoting vaginal health in adult woman reporting symptoms of vulvovaginal atrophy - VVA (or atrophic vulvovaginitis)

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged between 18 and 65 years.
2. Patients reporting vulvovaginal dryness associated with spontaneous pain and / or dyspareunia (minimum score of 30 on a 100 mm Visual Analogue Scale for both symptoms referable to vulvovaginal atrophy: dryness and spontaneous pain and / or dyspareunia).
3. Patients sexually active (i.e. women who currently have intercourse or other sexual activity (masturbation, etc) at least once a month (with or without a partner), or who had intercourse or other sexual activity at least once a month in the past, but later decreased sexual activity due to excessive pain or vaginal dryness. Dyspareunia is defined (2nd International Consultation on Sexual Medicine) as "persistent or recurrent pain with attempted or complete vaginal entry and/or penile vaginal intercourse" that is not the result of other abnormalities).
4. Patients agreeing not to use lubricants or other topically applied vaginal products during the study and not to modify their personal hygiene products.
5. Patients of childbearing potential following a reliable (according to investigator's opinion) non-hormonal contraception therapy.
6. Patients presenting body mass index between 18.5 and 29.9 kg/m2.
7. Patients with normal Papanicolaou test results (including inflammatory changes) within the past 12 months after specimen collection.
8. Willingness to participate in the study and to sign an informed consent form.
9. No past or present narcotic addiction or alcoholism.

Exclusion Criteria:

1. Patients presenting vulvar or vaginal pathology other than vulvovaginal atrophy.
2. Patients pregnant or breastfeeding.
3. Patients presenting undiagnosed abnormal genital bleeding.
4. Patients presenting endometrial pathology, such as hyperplasia (endometriosis) or endometrial polyps, cancer, palpable fibroids or grade 2 uterine prolapse (when the cervix reaches the labia minora) on gynaecologic examination.
5. Patients presenting coagulation disorders or on anticoagulant drug therapy (except clopidogrel or acetylsalicylic acid).
6. Patients diagnosed with clinically significant metabolic or endocrine disease or diabetes mellitus uncontrolled by medication.
7. Patients diagnosed with hypertension and in treatment with antihypertensive medications.
8. Patients diagnosed with severe renal and/or hepatic insufficiency.
9. Patients who have changed or started systemic oestrogen - progestin or hormone therapy in the 3 months prior to inclusion (including contraceptive therapy (pill) or Substitutive Hormonal Therapy (SHT)).
10. Patients on systemic chronic oestrogen - progestin therapy (including contraceptive therapy (pill) or Substitutive Hormonal Therapy (SHT)).
11. Patients in treatment with the following systemic drug: nonsteroidal anti-inflammatory drugs, antihistamines, corticosteroids in the 2 weeks prior to inclusion, immunosuppressants in the 3 months prior to inclusion, venotonic or diuretic agents in the month prior to inclusion.
12. Patients using topic oestrogen - progestin or hormonal therapy, in the week prior to inclusion.
13. Patients in treatment with topically applied vaginal products, including medications to promote healing, in the week prior to inclusion.
14. Patients that participated in any other clinical trial during the last month or participating in any clinical trial while participating in this trial.
15. Patients reporting allergy or intolerance to any component of test product, placebo or rescue product.
16. Smoking patients.
17. Patients who in the opinion of the principal investigator are at risk of non-compliance to the study procedures or who are otherwise not appropriate to include in this clinical trial.
18. Patients presenting contraindications to the rescue product, according to concerning Summary of Product Characteristics (SPC).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2019-09-24 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Assessment of Vaginal Health Index (VHI) | from Day 0 to Day 21
  comparison between groups, mean change from Day 0 to Day 21

SECONDARY OUTCOMES:
Assessment of vulvar signs of VVA assessed by means of vulvoscopy | from Day 0 to Day 21
  comparison between groups, mean change from Day 0 to Day 21
Assessment of vulvar signs of VVA (vaginal secretions, vaginal epithelial integrity, vaginal epithelial surface thickness and vaginal colour, categorized as none, mild, moderate, or severe corresponding to a score of 0, 1, 2 or 3, respectively) | from Day 0 to Day 21
  comparison between groups, mean change from Day 0 to Day 21
Assessment of visible skin signs of irritation such as redness, dryness, scaling, peeling, bumps, hives, categorized as none, mild, moderate, or severe corresponding to a score of 0, 1, 2 or 3, respectively | from Day 0 to Day 21
  comparison between groups, mean change from Day 0 to Day 21
Assessment done by Investigator of overall improvement by means of Global Assessment of Improvement (GAI - according to a 7-grade scoring system, 0-6) | at Day 21
  comparison between groups, at Day 21
Assessment of subjective vaginal symptoms related to VVA and irritation (dryness, dyspareunia, burning, itching, stinging) by means of 100 mm Visual Analogue Scales | from Day 0 to 21
  comparison between groups, mean change from Day 0 to Day 21
Assessment of global severity score for symptoms of VVA | from Day 0 to Day 21
  comparison between groups, mean change from Day 0 to Day 21
Assessment of dyspareunia by means of the Marinoff Dyspareunia Scale | from Day 0 to Day 21
  comparison between groups, mean change from Day 0 to Day 21
Assessment of pain through the short form of McGill Pain questionnaire | from Day 0 to Day 21
  comparison between groups, mean change from Day 0 to Day 21
Assessment of patient satisfaction, assessed on 0 to 10 points scale (extremely dissatisfied = 0; extremely satisfied = 10) | at Day 21
  comparison between groups, at Day 21
Patient willingness to use the product in the future, assessed on 1 - 4 points scale (strongly disagree=1, disagree=2, agree=3, strongly agree=4) | at Day 21
  comparison between groups, at Day 21
Assessment of rescue product use (starting date and number of times the rescue product was used) | at Day 21
  comparison among groups, at Day 21

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Spedali Civili di Brescia, Brescia
  - Istituto Europeo di Oncologia, Milan
  - Fondazione IRCCS Policlinico San Matteo, Pavia